CLINICAL TRIAL: NCT00363909
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Evaluation of Citalopram for the Treatment of Hot Flashes
Brief Title: Citalopram in Treating Postmenopausal Women With Hot Flashes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N05C9; NCI-2012-02699 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000489567 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer; Hot Flashes; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; hot flashes; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- low-dose citalopram hydrobromide (Experimental): Patients receive 1 tablet of oral citalopram once daily in weeks 2-7.
  All patients complete a diary of hot flash incidence in weeks 1-7 and undergo blood collection periodically during study treatment for translational research studies.
  Interventions: Drug: citalopram hydrobromide
- medium-dose citalopram hydrobromide (Experimental): Patients receive 1 tablet of oral citalopram once daily in week 2 and 2 tablets once daily in weeks 3-7.
  All patients complete a diary of hot flash incidence in weeks 1-7 and undergo blood collection periodically during study treatment for translational research studies.
  Interventions: Drug: citalopram hydrobromide
- high-dose citalopram hydrobromide (Experimental): Patients receive 1 tablet of oral citalopram once daily in week 2, 2 tablets once daily in week 3, and 3 tablets once daily in weeks 4-7.
  All patients complete a diary of hot flash incidence in weeks 1-7 and undergo blood collection periodically during study treatment for translational research studies.
  Interventions: Drug: citalopram hydrobromide
- placebo (Placebo Comparator): Patients receive 1-3 placebo tablets once daily in weeks 2-7.
  All patients complete a diary of hot flash incidence in weeks 1-7 and undergo blood collection periodically during study treatment for translational research studies.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: citalopram hydrobromide
  Arms: high-dose citalopram hydrobromide; low-dose citalopram hydrobromide; medium-dose citalopram hydrobromide
Other: placebo
  Arms: placebo

SUMMARY:
RATIONALE: Citalopram may help relieve hot flashes in women who had or have not had breast cancer. It is not yet known which dose of citalopram is more effective in treating hot flashes in postmenopausal women.

PURPOSE: This randomized phase III trial is studying three different doses of citalopram to compare how well they work in treating postmenopausal women with hot flashes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of three different doses of citalopram hydrobromide on hot flash scores in postmenopausal women with a history of breast cancer or in postmenopausal women who do not wish to take estrogen replacement therapy for fear of increased risk of breast cancer.

Secondary

* Compare the side effect profile of these regimens in these patients.
* Compare the effects of these regimens on the secondary outcome of mood and interference with activities from hot flashes.
* Determine if CYP2C19 and CYP2D6 polymorphisms predict efficacy of various doses of citalopram hydrobromide.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to age (18-49 years vs ≥ 50 years), tamoxifen (yes vs no), selective estrogen-receptor modulators (SERMs) (yes vs no), aromatase inhibitors (yes vs no), duration of hot flashes (< 9 months vs ≥ 9 months), and frequency of hot flashes per day (< 4 vs 4-9 vs ≥ 10). Patients are randomized to 1 of 4 treatment arms.

* Arm I (low-dose citalopram hydrobromide): Patients receive 1 tablet of oral citalopram once daily in weeks 2-7.
* Arm II (medium-dose citalopram hydrobromide): Patients receive 1 tablet of oral citalopram once daily in week 2 and 2 tablets once daily in weeks 3-7.
* Arm III (high-dose citalopram hydrobromide): Patients receive 1 tablet of oral citalopram once daily in week 2, 2 tablets once daily in week 3, and 3 tablets once daily in weeks 4-7.
* Arm IV (placebo): Patients receive 1-3 placebo tablets once daily in weeks 2-7. All patients complete a diary of hot flash incidence in weeks 1-7 and undergo blood collection periodically during study treatment for translational research studies.

A Symptom Experience diary is completed weekly and Profile of Mood States and Hot Flash-Related Interference Scale questionnaires are completed at baseline and in week 7.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must meet 1 of the following criteria:

  * History of breast cancer

    * No current malignant disease
  * No history of breast cancer and refused estrogen replacement therapy due to perceived increased risk of breast cancer
* Bothersome hot flashes, defined as hot flashes ≥ 14 times/week and of sufficient severity to make the patient desire therapeutic intervention
* Presence of hot flashes ≥ 1 month prior to study entry
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal, as defined by 1 of the following criteria:

  * Absence of a menstrual period in the past 12 months
  * Bilateral oophorectomy
  * Absence of a menstrual period in the past 6 months with follicle-stimulating hormone (FSH) level > 40 mIU/mL
* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* Willing to provide blood samples during study participation
* No history of allergic or other adverse reactions to citalopram hydrobromide or other selective serotonin reuptake inhibitors (SSRIs)
* No documented mania or hypomania

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior and no concurrent antineoplastic chemotherapy
* At least 4 weeks since prior and no concurrent androgens, estrogens, or progestational agents
* At least 3 months since prior antidepressant use, including Hypericum perforatum (St. John's wort)
* Concurrent tamoxifen, raloxifene, or aromatase inhibitors allowed if on a constant dose for ≥ 4 weeks and continuing medication during study period
* No other concurrent or planned agents for treating hot flashes (e.g., phenobarbital, megestrol, or clonidine)

  * Stable dose of vitamin E allowed as long as it was started > 30 days prior to study entry
* Concurrent soy allowed
* Concurrent gabapentin allowed for reasons other than hot flashes if on a constant dose for ≥ 1 month and continuing during study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2006-11; Primary Completion 2007-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Difference in average hot flash score from baseline until week 7 of treatment | Up to 7 weeks

SECONDARY OUTCOMES:
Toxicity | Up to 7 weeks
Mood- and hot flash-related daily interference with activities | Up to 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Debra Barton, RN, PhD, AOCN, FAAN, Study Chair — Mayo Clinic
Locations (198):
- United States (198):
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Immanuel St. Joseph's Clinic, Mankato, Minnesota
  - Minnesota Oncology Hematology, PA at Maplewood Cancer Center, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Hematology-Oncology Associates of Fredericksburg, Incorporated, Fredericksburg, Virginia
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Barton DL, LaVasseur BI, Sloan JA, Stawis AN, Flynn KA, Dyar M, Johnson DB, Atherton PJ, Diekmann B, Loprinzi CL. Phase III, placebo-controlled trial of three doses of citalopram for the treatment of hot flashes: NCCTG trial N05C9. J Clin Oncol. 2010 Jul 10;28(20):3278-83. doi: 10.1200/JCO.2009.26.6379. Epub 2010 May 24. PMID 20498389
- [Result] Barton DL, LaVasseur B, Sloan JA, et al.: A phase III trial evaluating three doses of citalopram for hot flashes: NCCTG trial N05C9. [Abstract] J Clin Oncol 26 (Suppl 15): A-9538, 2008.